CLINICAL TRIAL: NCT01713062
Title: Randomised Prospective Multicenter Longterm-Evaluation of the Survival Rate of the Implant, Wear and Periprosthetic Osteolysis of Highly Cross-linked Polyethylene With and Without Addition of Vitamin E (UHMWPE-XE vs. UHMWPE-X)
Brief Title: Longterm-Evaluation of Vitelene® Against Standard
Acronym: VITAS
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-G-H-1113
Record Dates: First submitted 2012-10-15; First posted 2012-10-24 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis, Hip; Arthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vitelene: Plasmacup DC® with Vitelene® inlay manufactured by UHMWPE-XE (Ultra High Molecular Weight Polyethylene highly cross-linked with 0.1% Vitamin E) in combination with one of four different Aesculap® stems (Bicontact®, TRJ®, Metha®, Excia®)
  Interventions: Device: Vitelene
- XLPE: Plasmacup DC® with a standard polyethylene inlay manufactured by UHMWPE-X (Ultra High Molecular Weight Polyethylene highly cross-linked) in combination with one of four different Aesculap® stems (Bicontact®, TRJ®, Metha®, Excia®)
  Interventions: Device: XLPE

INTERVENTIONS:
Device: Vitelene — THA
  Groups: Vitelene
Device: XLPE — THA
  Groups: XLPE

SUMMARY:
The purpose of this randomised prospective multicenter longterm study is to evaluate the survival rate of the implant, wear and periprosthetic osteolysis of highly cross-linked polyethylene with and without addition of Vitamin E (UHMWPE-XE vs. UHMWPE-X) in Total Hip Arthroplasty.

ELIGIBILITY:
Inclusion:

* Minimum age: 18 years
* Maximum age: 75 years
* Indication of cementless THA
* Approval of study participation and treatment according to study protocol
* Physical and mental willingness of adhering to clinical and radiological follow up

Exclusion:

* Patient is not able to join follow up
* Increased risk of anaesthesia according to the "American Society of Anesthesiology": ASA IV
* Tumor disease
* Alcohol and drug dependency
* Permanent cortisone therapy
* Clinical relevant infections
* Pregnancy and planned pregnancy
* Previous interventions like adjustment-osteotomy, treatment of fractures or THA on affected side
* Acute fractures of the affected hip joint
* Patients with bone quality, which doesn´t allow a cementless treatment
* Requirements of clinical relevant deformities (condition after preoperation or bone fracture, leg length discrepancy > 30 mm, Offset-reduction about > 30 mm)
* Small acetabular treatments with 28 mm heads
* Treatments without using ceramic heads
* Treatments which require neck prolonging components

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Analysis and measurement of oxidation index of the Polyethylene Inlay after Revision | Oxidation index is assessed in case of loosening and revision within 15 years
  The Oxidation index is measured after explantation in case of loosening of the inlay

SECONDARY OUTCOMES:
Manifest radiological osteolyses | Measured radiologically after 1, 5, 10 and 15 years
Traceable wear of polyethylene over 0.5 mm | Measured radiologically after 1, 5, 10 and 15 years
Clinical Outcome | After 1, 5, 10 and 15 years
  Clinical Outcome measured by Harris Hip Score (HHS), Hip disability and osteoarthritis outcome score(HOOS), University of California at Los Angeles Score (UCLA)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Jäger, Prof. Dr. med, Principal Investigator — Universitätsklinikum Essen
Locations (6):
- Germany (6):
  - Fachklinik für Orthopädie, Unfallchirurgie, WirbelsäulenchirurgieMarienhaus Klinikum St. Josef, Bendorf
  - Klinik für Orthopädie und Unfallchirurgie, Bochum
  - Klinik und Poliklinik für Orthopädie, Halle
  - Orthopädische Klinik der MHH im Annastift, Hanover
  - St. Marien Hospital, Mülheim
  - Elisabeth Klinikum Olsberg, Olsberg